CLINICAL TRIAL: NCT05797649
Title: Comparing N-terminal-proB-type Natriuretic Peptide with Other Diagnostic Criteria in Discriminating Heart Failure-associated from Non-heart Failure-associated Pleural Effusions
Brief Title: Comparing the Diagnostic Sensitivity and Specificity of Pleural Fluid N-Terminal Pro B-type Natriuretic Peptide (NT-proBNP) and Other Biochemical Gradient Criteria in Distinguishing Heart Failure and Non-heart Failure Related Pleural Effusions (CENTRE Study)
Status: Recruiting | Type: Observational
Sponsor: Chinese University of Hong Kong (Other)
Collaborators: Roche Diagnostics GmbH (Industry)
Responsible Party: Principal Investigator, Christopher Chan, Honorary Clinical Tutor, Chinese University of Hong Kong
Other Study IDs: NTProBNPPleuralEffusion1
Record Dates: First submitted 2023-03-16; First posted 2023-04-04 (Actual); Last update posted 2024-11-13 (Actual); Status verified 2024-11

CONDITIONS: Pleural Effusion; Heart Failure; Malignant Neoplasm; Fluid Overload; Hypoalbuminemia; Renal Failure; Cirrhosis; Infections
Keywords: pleural fluid; heart failure; malignancy; cancer; echocardiography; infection; tuberculosis; respiratory medicine
MeSH Terms: conditions — Pleural Effusion; Heart Failure; Neoplasms; Edema; Hypoalbuminemia; Renal Insufficiency; Fibrosis; Infections; Tuberculosis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 24 Months
Biospecimen Retention: Samples Without DNA — Pleural Fluid and Blood
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Heart Failure-Associated Pleural Effusion: Patients with pleural effusion with an underlying aetiology of heart failure
- Control group: Patients with pleural effusion due to exudative, or non-fluid overload causes

SUMMARY:
To assess the discriminative properties of pleural fluid (PF) N-terminal-proB-type-natriuretic-peptide (NTproBNP) levels in identifying heart failure (HF)-associated pleural effusions (PE).

DETAILED DESCRIPTION:
Objective: To assess the discriminative properties of pleural fluid (PF) N-terminal-proB-type-natriuretic-peptide (NTproBNP) levels in identifying heart failure (HF)-associated pleural effusions (PE).

Hypothesis to be tested: The PF NTproBNP levels are superior to existing methods including Light's criteria, serum/pleural fluid (S/PF) protein gradient, and albumin gradient, in identifying transudates and distinguishing between HF- and non-HF-associated PE.

Design and subjects: A prospective case-control study involving patients with PE requiring thoracentesis, caused by hypervolaemia due to HF, diseases other than HF, and patients with pleural effusion without hypervolaemia. Patient characteristics, PF results and effusion aetiology will be analysed. Patient outcomes will be followed up to 3 months to confirm the aetiology of PE. Clinical management of patients will not be affected.

Study instruments: PF of recruited patients will be analysed for albumin, protein, lactate dehydrogenase (LDH) levels and NTproBNP. The diagnosis of HF will be based on clinical features, serum NTproBNP and echocardiogram.

Main outcome measures: The performance of PF NTproBNP level in identifying HF-associated PE.

Data analysis: The PF NTproBNP level will be compared between effusions of different aetiologies. The optimal pleural fluid NTproBNP level with largest area under the receiver operating characteristic curve in identifying HF-associated PE will be determined. Performance of PF NTproBNP level in identifying HF-associated PE, and other biochemical criteria in identifying transudates will be compared. Echocardiographic findings will be correlated with the PF NTproBNP levels.

Expected results: The diagnostic performance of PF NTproBNP will be significantly better in identifying HF-associated effusion than other biochemical criteria.

ELIGIBILITY:
Inclusion Criteria:

* Patients hospitalized for heart failure and pleural effusion
* Pleural tapping indicated for pleural fluid analysis.
* Aged 18 years old or above

Exclusion Criteria:

* History of intrapleural therapy (including talc and fibrinolytic) in the ipsilateral pleural space.
* History of surgical decortication or pleurodesis in the ipsilateral pleural space.
* Ipsilateral thoracic or cardiac surgery in the past 3 months.
* Failure to obtain informed consent due to the patient's refusal or cognitive impairment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who are admitted to the Department of Medicine & Therapeutics, Prince of Wales Hospital (PWH) who fulfil the inclusion and exclusion criteria
Sampling Method: Non-Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2023-07-01 (Actual); Primary Completion 2025-11-30 (Estimated); Study Completion 2025-11-30 (Estimated)

PRIMARY OUTCOMES:
Comparison of the diagnostic performance of PF NTproBNP level in the diagnosis of HF-associated pleural effusions with other conventional biochemical criteria | 24 months
  Pleural fluid NTproBNP will be measured in patients with pleural effusion of various aetiologies including malignancy, pleural infection, heart failure and other causes of volume overload. The sensitivity and specificity of an elevated pleural fluid NTproBNP level in successfully identifying a pleural effusion due to underlying heart failure will be measured and compared against existing classification criteria for pleural effusion such as Light's Criteria, pleural-serum protein gradient or albumin gradient.

SECONDARY OUTCOMES:
To measure the PF NTproBNP level in patients with pleural effusion of various aetiologies | 24 months
Correlation of clinical factors that may affect the levels of pleural fluid NTproBNP such as echocardiographic features, presence of comorbidities, nutritional status, serum albumin level, levels of inflammatory markers and presence of infection | 24 months
  Clinical data of patients admitted to the hospital with pleural effusion will be measured and recorded. Statistical analysis will then be performed to evaluate for degree of correlation between the presence or severity of a clinical parameter, echocardiogram results e.g. severe valvular stenosis, or, e.g. presence of medical comorbidities or presence of concomitant infection, and the levels of NTproBNP identified in the patient's pleural fluid detected within same admission.
To correlate the PF NTproBNP levels with the echocardiographic features and prognosis of patients with heart failure | 24 months

CONTACTS AND LOCATIONS:
Locations (1):
- Prince of Wales Hospital, Hong Kong, New Territories, Hong Kong

IPD SHARING:
Plan to Share IPD: No
Given patient data and privacy concerns, clinical data involving individual patients will not be shared. Data summary tables may later be published along with the research manuscript, and may be shared upon receipt of a reasonable request.